CLINICAL TRIAL: NCT04869891
Title: How Much The Self-Reported Physical Activity Change in Patients With Physical Disabilities Hospitalized for Rehabilitation in A Physical Medicine and Rehabilitation Clinic
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Damla Cankurtaran, Medical doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: PASIPD
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Disability Physical; Impairment; Physical Activity; Rehabilitation; Televisit
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Disability was defined by WHOas a restriction or lack of ability to perform daily activity, but this definition was later changedto problems in functioning in the WHO classification of Functioning, Disability and Health (ICF). Osteoarthritis, back pain, neck pain, rheumatologic diseases, neurologic disorders (stroke, spinal cord injury, multiple sclerosis, Parkinson diseases) can cause physical disabilities.Recent studies have shown that; high levels ofdisability is related with low levels of physical activity.Individuals with disability are commonly hospitalized ininpatients clinicsfor rehabilitation, which aims to achieveoptimal functional level ofpatients within their own limitations.A rehabilitation program can be an excellent opportunity to integrate post-rehabilitation physical activity into their lifestyle.This study aimed to examine the short term effect of inpatient rehabilitation program on self -reported physical activity both participants with physical disabilities due to musculoskeletal, and neurological disorders

ELIGIBILITY:
Inclusion Criteria:

* Patients with physical disabilities, due to neurologic or musculoskeletal diseases and hospitalized in PMR clinic for rehabilitation between Patients over 18 years of age with cognitive functions able to fill the forms and patients with medical stabilization for neurological diseases.

Exclusion Criteria:

* Patients under 18 years of age,
* Patients with additional hearing, visual and mental disabilities
* Patients with metabolic instability for neurological diseases, history of malignancyand pulmonary and cardiac failure,
* Patients with recurrent hospitalization in the PMRclinic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with physical disabilities, due to neurologic or musculoskeletal diseases and hospitalized in PMR clinic for rehabilitationbetween September 2020 andMarch 2021were
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
PASIPD | 15 MİNUTES
  SELF-REPORTED PHYSİCAL ACTİVİTY

CONTACTS AND LOCATIONS:
Locations (1):
- DiskapiYBERH, Çankaya, Ankara, Turkey (Türkiye)